CLINICAL TRIAL: NCT02785640
Title: A Study to Assess the Impact of a Multicomponent Intervention to Reduce Prolonged Sitting in the Workplace
Brief Title: Prompting Activity in a Workplace Setting
Acronym: PAWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GlasgowCU2
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prompt group (Experimental): Following feedback on their baseline sitting behaviour and an education session on the health benefits of breaking prolonged sitting, the prompt group will receive hourly prompts on their PC to stand. The prompts will be delivered via Microsoft Outlook and will run for a period of 10 weeks. The messages will be short in length, varied and centre around the key message of breaking prolonged sitting by standing
  Interventions: Behavioral: Hourly prompts to stand delivered by Microsoft Outlook
- Control group (No Intervention): The control group will receive the same education session as the prompt group, as well as feedback on their baseline sitting behaviour. However, the will not receive prompts on their PC.

INTERVENTIONS:
Behavioral: Hourly prompts to stand delivered by Microsoft Outlook — Prompt group
  Arms: Prompt group

SUMMARY:
This dual-arm randomised study aims to test a multi-component intervention to reduce sedentary behaviour in a cohort of desk-based office workers.

DETAILED DESCRIPTION:
There is increasing evidence to demonstrate that excessive and unhealthy patterns of sedentary behaviour can increase the risk of a range of health problems,independent to levels of physical activity. Increasingly, people are employed in low activity occupations with office workers being identified as one of the most sedentary roles. Small scale studies using prompts to remind office workers to stand have shown promising results, as well as representing a low-cost solution for employers. This study builds upon a recent pilot study investigating the impact of prompts delivered via Microsoft Outlook, on the sedentary behaviour of office workers.

Developed in accordance with the Medical Research Council framework for designing multi-component interventions this study utilises Social Cognitive Theory (SCT) as a theoretical basis. SCT describes the complex interaction between individuals and their environment. The influence of the office environment on sedentary behaviour is clearly illustrated by differences in people's sitting patterns inside and outside of working hours . Behavioural change techniques linked to the constructs of SCT have also been shown to have a positive impact on sedentary behaviour, namely education, goal setting and feedback. Participants in this study will therefore receive education on the benefits of breaking their sitting, tips on how to achieve this, and feedback on their baseline sitting behaviour. This study will test the impact of these techniques on sitting time and patterns, and also track their influence on the different constructs of SCT and individuals' readiness to change by measuring these at time points throughout the intervention. To address the fact that sitting at work may not be a conscious decision, but performed out of habit, half of participants will also receive prompts reminding them to stand. The same prompts will be used as in the pilot study, but the addition of an extra activity monitoring period will enable us to ascertain whether the impact of prompts diminishes during the intervention period.

This study will aim to recruit 60 desk-based office employees via email invitation. Volunteers will be screened using inclusion/exclusion criteria and asked to provide signed consent. Sitting will be de-emphasised in the participant information sheet, and other documentation used at recruitment, in order to minimise any impact on baseline activity measurements. Cluster randomisation will be used to split participants into two equal groups (Group 1 n=30, group 2 n=30) based on their physical location within the office(s) in order to minimise contamination between groups. Randomisation software will be used to allocate groups on www.randomisation.com. Baseline measurement for all participants will consist of completion of questionnaires and activity monitoring as follows:

1. Questionnaires:

   * Q1: Demographic data - to obtain basic information on participants
   * Q2: Stage of change questionnaire - measuring readiness to change
   * Q3: Social cognitive theory questionnaire - measuring key constructs of SCT
2. Activity monitoring:

   * Participants will be asked to wear a water-proofed activPAL activity monitor* on the front of their thigh for a period of 7 consecutive days (24 hours a day)
   * A brief diary will be completed for the same 7 days

     * The activPAL activity monitor has been validated for measuring and categorising sitting/lying, standing and walking using an acceleration signal from the thigh .

Following the collection of baseline data, all participants will attend a 1 hour education session during which they will receive a presentation outlining: the health problems associated with prolonged sedentary behaviour; how much sitting is recommended; feedback on their own baseline sitting behaviour; and tips on how to reduce and break up sedentary behaviour. They will be given a summary of their baseline activity data . Group 1 will then return to work as normal. Group 2 will receive an excel file to upload to Microsoft Outlook which will deliver prompts to break sitting at random times, once within an hour. The prompts will run for a period of 10 weeks and their content will be the same brief, positively framed messages that were evaluated favourably by participants in the pilot project. Measurements for all participants will be repeated as follows: Questionnaires Q2 and Q3 will be repeated after the education session and at 12 week follow-up; 1 week of activity monitoring will be repeated between weeks 2-4 of the intervention period, 8-10 of the intervention period, and at 12 week follow up.

Following final measurements, participants will be invited to one of a series of semi-structured focus groups to explore the feasibility, acceptability, meaningfulness and effectiveness of the intervention. Focus groups will be recorded using a digital voice recorder and transcribed.

Data will be treated as confidential, it will be anonymised, and stored securely in line with GCU's data protection policies. Electronic copies of the activity data will be kept for 10 years, alongside electronic and paper copies of the questionnaires and diaries and audio and transcribed accounts of the focus groups. Physical activity data and basic demographic data will also be kept on a password protected database on a secure server. The data held on the database will not be identifiable. The information collected may be used for further analysis by staff and students in the School of Health and Life Sciences at Glasgow Caledonian University at a later date. Access to data will be restricted and controlled by Dr Ben Stansfield, PGRT in the School of Health and Life Sciences, GCU. Individuals will not be identifiable from any reports published and the employer, JJML, will receive a report containing only amalgamated data.

: Each participant will receive a brief summary of their baseline activity data at the education session. In addition, at the end of the study they will be provided with an activity report, summarising their individual activity data for all 4 measurement periods. A report of amalgamated data, including the results of the focus groups, will be produced for JJML and this will also be made available to study participants. Furthermore, the results will be written up as a PhD thesis, published in appropriate academic journals and discussed in conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Primarily engaged in sedentary, computer-based activities
* Access to Microsoft Outlook calendar

Exclusion Criteria:

* Workstation comprises of a standing desk
* Pre-existing health condition that prevents standing on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total time spent sitting at work | 12 weeks
  Total time spent sitting at work will be objectively measured using a tri-axial accelerometer

SECONDARY OUTCOMES:
Total time spent sitting at work in continuous bouts of at least 30 minutes. | 12 weeks
  This will be objectively measured using a tri-axial accelerometer
Number of sitting events at work | 12 weeks
  These will be objectively measured using a tri-axial accelerometer
Number of prolonged sitting events at work | 12 weeks
  Number of sitting events that last at least 30 minutes at work will be objectively measured using a tri-axial accelerometer
Time after prompt to stand | 12 weeks
  The amount of time it takes those in the intervention group to stand following delivery of a prompt will be objectively measured using a tri-axial accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Dall, PhD, Principal Investigator — Senior Research Fellow
Locations (1):
- Glasgow Caledonian University, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chau JY, Grunseit AC, Chey T, Stamatakis E, Brown WJ, Matthews CE, Bauman AE, van der Ploeg HP. Daily sitting time and all-cause mortality: a meta-analysis. PLoS One. 2013 Nov 13;8(11):e80000. doi: 10.1371/journal.pone.0080000. eCollection 2013. PMID 24236168
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Background] Owen N, Healy GN, Matthews CE, Dunstan DW. Too much sitting: the population health science of sedentary behavior. Exerc Sport Sci Rev. 2010 Jul;38(3):105-13. doi: 10.1097/JES.0b013e3181e373a2. PMID 20577058
- [Background] Parry S, Straker L, Gilson ND, Smith AJ. Participatory workplace interventions can reduce sedentary time for office workers--a randomised controlled trial. PLoS One. 2013 Nov 12;8(11):e78957. doi: 10.1371/journal.pone.0078957. eCollection 2013. PMID 24265734
- [Background] Healy GN, Lawler S, Thorp A, Neuhaus M, Robson E, Owen N, et al. Reducing prolonged sitting in the workplace. An evidence review: full report. 2012;ISBN:978-1-921822-06-3.
- [Background] Evans RE, Fawole HO, Sheriff SA, Dall PM, Grant PM, Ryan CG. Point-of-choice prompts to reduce sitting time at work: a randomized trial. Am J Prev Med. 2012 Sep;43(3):293-7. doi: 10.1016/j.amepre.2012.05.010. PMID 22898122
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Bandura A, 1925. Self-efficacy: the exercise of control / Albert Bandura. New York: W.H. Freeman; 1997.
- [Background] Gardner B, Smith L, Lorencatto F, Hamer M, Biddle SJ. How to reduce sitting time? A review of behaviour change strategies used in sedentary behaviour reduction interventions among adults. Health Psychol Rev. 2016;10(1):89-112. doi: 10.1080/17437199.2015.1082146. Epub 2015 Sep 16. PMID 26315814
- [Background] Neuhaus M, Healy GN, Dunstan DW, Owen N, Eakin EG. Workplace sitting and height-adjustable workstations: a randomized controlled trial. Am J Prev Med. 2014 Jan;46(1):30-40. doi: 10.1016/j.amepre.2013.09.009. PMID 24355669
- [Background] Healy GN, Eakin EG, Lamontagne AD, Owen N, Winkler EA, Wiesner G, Gunning L, Neuhaus M, Lawler S, Fjeldsoe BS, Dunstan DW. Reducing sitting time in office workers: short-term efficacy of a multicomponent intervention. Prev Med. 2013 Jul;57(1):43-8. doi: 10.1016/j.ypmed.2013.04.004. Epub 2013 Apr 15. PMID 23597658
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Cooley D, Pedersen S. A pilot study of increasing nonpurposeful movement breaks at work as a means of reducing prolonged sitting. J Environ Public Health. 2013;2013:128376. doi: 10.1155/2013/128376. Epub 2013 Apr 3. PMID 23690798
- [Background] Grant PM, Ryan CG, Tigbe WW, Granat MH. The validation of a novel activity monitor in the measurement of posture and motion during everyday activities. Br J Sports Med. 2006 Dec;40(12):992-7. doi: 10.1136/bjsm.2006.030262. Epub 2006 Sep 15. PMID 16980531